CLINICAL TRIAL: NCT03432078
Title: Comparison of Effects Between Gut Directed Hypnotherapy Provided Either Individually or in a Group Setting for Patients With Irritable Bowel Syndrome (IBS) a Randomized Controlled Study.
Brief Title: Individual vs. Group Hypnotherapy in Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 686-11
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual hypnotherapy (Active Comparator): Treatment given on a individual basis, face to face.
  Interventions: Other: Hypnotherapy
- Group hypnotherapy (Active Comparator): Treatment given in a group setting, face to face.
  Interventions: Other: Hypnotherapy

INTERVENTIONS:
Other: Hypnotherapy — Non-pharmacological treatment

SUMMARY:
Patients' fulfilling Rome III criteria for IBS with symptoms refractory to standard treatment who are referred to a specialist unit for hypnotherapy are consecutively included in the study. The patients are randomized to either individual or group treatment given by a nurse trained in hypnotherapy. The treatment consists of eight sessions of gut directed hypno therapy during twelve weeks. Effects are measured by validated questionnaires at baseline and at various time points during the treatment period as well as after the completion of the treatment.

DETAILED DESCRIPTION:
Patients' fulfilling Rome III criteria for IBS with symptoms refractory to standard treatment who are referred to a specialist unit for hypnotherapy are consecutively included in the study. Firstly, the patients are invited to a meeting with the nurse for information about the study, check for eligibility and to sign the written informed consent. Exclusion criteria that could influence GI symptoms such as organic GI disease, severe psychiatric comorbidity and pregnancy are controlled for. The patients are randomized to either individual or group treatment given by a nurse trained in hypnotherapy and cognitive behavioral therapy. The randomization is organized and performed in blocks by an external unit connected to the University in order to be accurate. The treatment consists of eight sessions of gut directed hypnotherapy during twelve weeks. A standardized protocol is used and is the same both in the group setting as well as in the individual treatment arm. In each group approximately eight patients are included. Every session lasts for one hour. Outcome measures in the study are GI symptom severity, GI-specific anxiety, psychological distress and health related quality of life. These effects are measured by validated questionnaires at baseline and at various time points during the treatment period as well as after the completion of the treatment and during the 6 months-, 1 and 2 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to Rome III criteria

Exclusion Criteria:

* Organic GI disease

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Gastrointestinal symptom severity | Up to ten years
  Measured with Irritable Bowel Syndrome- severity scoring system (IBS-SSS). The questionnaire measures severity of GI symptoms and consists of five questions where each score ranges from 0 to 100. A total score of all five questions is calculated ranging from 0 to 500. The higher the score the more severe the GI symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovdahl J, Blomqvist-Storm M, Palsson OS, Ringstrom G, Tornblom H, Simren M, Trindade IA. Nurse-Administered Gut-Directed Hypnotherapy for Irritable Bowel Syndrome: A Two-Year Follow-Up Study. United European Gastroenterol J. 2025 Sep;13(7):1307-1317. doi: 10.1002/ueg2.70060. Epub 2025 Jun 9. PMID 40491242
- [Derived] Lovdahl J, Tornblom H, Ringstrom G, Palsson OS, Simren M. Randomised clinical trial: individual versus group hypnotherapy for irritable bowel syndrome. Aliment Pharmacol Ther. 2022 Jun;55(12):1501-1511. doi: 10.1111/apt.16934. Epub 2022 May 3. PMID 35505463